CLINICAL TRIAL: NCT04753593
Title: Use of Discarded Surgery Human Tissue Specimens for Basic Science Research
Acronym: HumTisRes
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0002
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Osteoblast; Vascular Calcification
Keywords: osteoblast; Vascular Calcification; vascular smooth muscle cell; Cardiac valve calcification; Valvular interstitial cell; bone tissue
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — discarded human tissue fragments : vessel and bone tissue that are been harvested during surgery and which are not intended to be used for clinical-biological management of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although it is now established that calcification process result from the joint and coordinated action of different cell types, many areas of shadow remain regarding the spatio-temporal implementation of these events. Highlighting these processes requires additional research to consider new approaches to clinical management of patients with such conditions. It is in this context that the investigators need to use residual human tissue fragments resulting from surgery which are not intended to be used for clinical-biological management of patients. The use of these pseudonymised human tissues will allow the investigators to conduct in vitro cell culture experiences.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery in the Cardiac Surgery and Orthopedic Surgery departments of the CHU Amiens-Picardie
* patients who will be beforehand informed
* patients who will not be opposed to this study.

Exclusion Criteria:

* HIV and hepatitis positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aortic wall and aortic valve discarded specimens will come from the Cardiac Surgery department of Amiens Picardie CHU. The bone and peri-bone discarded specimens will come from the orthopedic surgery services of the CHU Amiens-Picardie.
  The collection of samples and their use is part of various projects carried out by research project leaders supported by the laboratory MP3CV (CURS, site CHU sud, Amiens). No genomic analysis is planned for these samples. None clinical data is associated with the interpretation of data collected through the work that will be carried out from these human tissue samples. There are no collections per se, the samples collected are pseudonymized.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Success in establishment of Cell Culture Systems from discarded surgery specimens | 5 years
  Success in establishment of Cell Culture Systems from discarded surgery specimens

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France